CLINICAL TRIAL: NCT05230446
Title: PRospective Evaluation of Complete Revascularization in Patients With multiveSsel Disease Excluding chroNic Total Occlusions
Acronym: PRESENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Roberto Diletti, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76556.078.21
Record Dates: First submitted 2021-11-23; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Multi Vessel Coronary Artery Disease; Non-ST Elevation Myocardial Infarction; Unstable Angina; Stable Angina; Coronary Artery Disease; Percutaneous Coronary Intervention; Optical Coherence Tomography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable; Angina, Stable; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous Coronary Intervention (Other): Interventional comparitor, compared to an optimal performance goal of 7% MACCE resulted from past CABG results
  Interventions: Device: PCI with OCT guidance

INTERVENTIONS:
Device: PCI with OCT guidance — Procedure will be optimize using pre-and post-stent OCT imaging, to improve the accuracy of stent placement and reduce geographic miss, but also to prevent malapposition of the stent and to discover dissections.

SUMMARY:
This prospective, multicenter, non-randomized, single arm, objective performance goal (OPG) study is designed to evaluate clinical outcomes after complete revascularization by PCI and imaging guidance (OCT) in patients with multivessel coronary artery disease including left anterior descending (LAD) presenting with stable angina, or documented silent ischemia, or non-ST segment elevation acute coronary syndrome (NSTE-ACS).

DETAILED DESCRIPTION:
The PRESENT is an investigator-initiated, prospective, multicenter, non-randomized, single arm, OPG study. The objective performance goal is based on past results of CABG namely a rate of 7% MACCE at 1-year follow-up. All patients with multivessel disease without chronic total occlusion (CTO) and accepted for PCI are eligible for inclusion

Primary endpoint The primary clinical endpoint of this study is a composite of death from any cause, stroke, myocardial infarction, or unplanned ischemia driven repeat revascularization at 1-year post index procedure.

Secondary endpoint

* Composite of death from any cause, stroke, myocardial infarction, or repeat revascularization at 30 days, 2, and 5 years post intervention.
* All-cause mortality at 30 days, 1, 2, and 5 years
* Myocardial Infarction at 30 days, 1, 2, and 5 years
* Any revascularization at 30 days, 1, 2, and 5 years
* Stroke at 30 days, 1, 2, and 5 years
* Major bleeding at 30 days and 12 months
* Need for renal replacement therapy at 30 days

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, ≤85 years
2. The patient is an acceptable candidate for treatment with a drug eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, manufacturer's Instructions for Use and the Declaration of Helsinki
3. Patient indication, lesion length and vessel diameter of the target lesion(s) are according to the 'Instructions for Use' that comes with every Resolute Onyx (Zotarolimus-Eluting stent) system.
4. The patient is willing and able to cooperate with study procedures and required follow up visits
5. The subject or legal representative has been informed of the nature of the study and agrees to its provisions and has provided an EC approved written informed consent, including data privacy authorization

Exclusion Criteria:

1. Age <18 years and > 85 years.
2. Single coronary vessel disease.
3. No left anterior descending lesion.
4. Patients in cardiogenic shock.
5. Patients with STEMI.
6. Presence of a chronic total occlusion (CTO) defined as coronary lesion with Thrombolysis in Myocardial Infarction (TIMI) flow grade 0 on initial angiography present for more than or equal to 3 months.
7. Left main coronary artery disease
8. Patients who cannot give informed consent or have a life expectancy of less than 12 months.
9. Absolute contraindications or allergy that cannot be pre-medicated, to iodinated contrast or to any of the study medications, including both aspirin and P2Y12 inhibitors.
10. Patients with an extreme LAD tortuosity imparing OCT catheter advancement
11. Enrollment in another study with another investigational device or drug trial that has not reached the primary endpoint. The patient may only be enrolled once in the PRESENT study.
12. Previous coronary artery bypass grafting (CABG).
13. Patient requiring additional cardiac surgery within 6 months.
14. Women of childbearing potential who do not have a negative pregnancy test result within 7 days before the procedure, women who are known to be pregnant, or who are breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-11-18 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
MACCE- 1 year | 1 year
  The primary clinical endpoint of this study is a composite of death from any cause, stroke, myocardial infarction, or unplanned ischemia driven repeat revascularization at 1-year post index procedure.

SECONDARY OUTCOMES:
MACCE | 30 days, 2, and 5 years post intervention
  Composite of death from any cause, stroke, myocardial infarction, or repeat revascularization
All-cause mortality | 30 days, 1, 2, and 5 years
  All-cause mortality
Myocardial Infarction | 30 days, 1, 2, and 5 years
  Myocardial Infarction
Any revascularization | 30 days, 1, 2, and 5 years
  Any revascularization
Stroke | 30 days, 1, 2, and 5 years
  Stroke
Major bleeding | 30 days and 12 months
  Major bleeding according to the ARC criteria
Renal replacement therapy | 30 days
  Need for renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Diletti, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands